CLINICAL TRIAL: NCT06811181
Title: Study of Psychosocial and Contextual Determinants of General Practitioners' Management of Burnout
Acronym: BOPEC-MG
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Angers University Hospital (Unknown); National Research Agency, France (Other); IGEIA, audit intervention formation recherche en santé, F-44000 Nantes, France (Unknown); Tours university (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC24_0566
Record Dates: First submitted 2025-01-30; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Burnout
Keywords: Burnout; primary care; general practitioners
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General practitioners: Only practising French GPs will be included in the study. In qualitative phase, each GP will be interviewed during a research interview lasting one to one-and-a-half hours. In quantitative phase, GPs will receive an e-mail with a link to complete the questionnaire. The survey will take 15 minutes to complete.
  For the inclusion of participants in the qualitative phase, the sampling method chosen is that of maximum variation. The criteria used are: gender, age, seniority, type of agreement, type of territory, type of work organization.
  The quantitative phase involves sending a questionnaire by email to a professional mailing list of general practitioners.

SUMMARY:
Burnout is a major public and occupational health issue. Despite accumulated knowledge to date on the determinants of burnout and its treatment, shortcomings when providing support against this complex phenomenon have been found. Although many professionals are involved in the management of burnout, general practitioners (GPs), as primary care providers, are on the front line, and face a range of difficulties that are reflected in the wide variability of medical support brought to the patients. As a result, the diversity of these practices can affect the recovery process of burnout sufferers and their ability to return to work. Deviations from recommended practices can lead to shortcomings in the treatment of burnout. Using an exploratory et descriptive study design, the main objective of BOPEC-MG is to describe the psychosocial mechanisms involved in the management of burnout in general practice that could explain the variation in medical practices.

DETAILED DESCRIPTION:
The principal aim of this interdisciplinary project is to conduct an exploratory study of GPs' attitudes, beliefs and social representations with regard to burnout management, in order to better understand how their perceptions of this syndrome can influence their practices.

A mixed method combining qualitative and quantitative data collection will be used with samples from the French GPs population.

In phase 1 (qualitative study), semi-structured interviews will be conducted to explore:

1. The contextual aspects of professional practice (e.g. barriers to work);
2. The attitudes, beliefs and social representations about burnout;
3. Concrete practices for managing burnout (e.g. prescribing sick leave).

In addition to semi-structured interviews, qualitative data collection will include the examination of fictional clinical cases to describe medical practices. The format of the four fictional will be video, with actors playing the roles of patients with severe burnout in general practice. The independent variables manipuled will be age and gender.

In phase 2 (quantitative study), a questionnaire will be sent to french general practitioners. it will include scales developed using the results of phase 1 and scales validated by the scientific literature.

As for quantitative data collection, in addition to scales dedicated to attitudes, beliefs and practices, a questionnaire will include a free association task to describe social representations of burnout.

the questionnaire will measure:

1. attitudes
2. beliefs
3. social representations
4. screening for burnout and depression
5. contextual and environmental psychosocial determinants
6. care practices
7. socio-demographic variables

A randomized controlled trial aimed at harmonizing practices in general practice could be carried out on the basis of the results. Furthermore, the applications of the present study will be twofold: designing training courses in burnout management for the medical population, and contributing to communication campaigns to encourage GPs to follow the recommendations.

ELIGIBILITY:
Inclusion Criteria:

* practicing GPs
* GPs in northwestern region of France
* GPs with regular use of sick leave prescriptions

Exclusion Criteria:

* GPs with particular mode of exercise (e.g. 100% homeopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active general practitioners in the northwestern of France (around 23000 GPs)
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Attitudes and beliefs about burnout will be assessed with scales developed specifically on the basis of the qualitative results. | 1 day. Each participant is assessed one time
  Attitude and belief scales will include a series of items and statements relating to burnout and its management. The measurement method chosen is the Lickert scale, classically used for attitude assessment.
  The items and statements will be based on the content of the interviews (qualitative phase). The items will be subjected to a 3-stage judges' validation test:
  1. written judgment on each item,
  2. perfect agreement by the judges as to the unfavorable or favorable value of an item,
  3. 3 out of 4 judges agree that the statement is an attitude or belief. The items selected by this method will constitute the first operational version of the scale.

SECONDARY OUTCOMES:
Social representations about burnout will will be assessed with a free association test (Vergès, Scanon & Junique, 2005). | 1 day. Each participant is assessed one time
  The free association task is the method traditionally used to measure social representations. It consists in proposing an inductive word and asking the participant to evoke the 5 words related to this inductive term. This procedure has the advantage of being quick and encouraging spontaneity, which favors less controlled responses than in a qualitative survey. (Guimelli & Abric, 2007).
  In the context of this research, the inducer words will be: "burnout", "sick leave", "general practitioner".

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No